CLINICAL TRIAL: NCT03520010
Title: A Cluster Randomized Trial to Assess the Impact of Facilitated Implementation on Antibiotic Stewardship in Wisconsin Nursing Homes
Brief Title: Facilitated Implementation of Antibiotic Stewardship in Wisconsin Nursing Homes
Acronym: IMUNIFI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2018-0125; A534265 (Other: UW Madison); SMPH/MEDICINE/MEDICINE*I (Other: UW Madison); Protocol Version 6/16/2020 (Other: UW Madison)
Record Dates: First submitted 2018-04-26; First posted 2018-05-09 (Actual); Last update posted 2021-12-23 (Actual); Status verified 2021-12

CONDITIONS: UTI - Urinary Tract Infection
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internally-driven implementation (Active Comparator)
  Interventions: Behavioral: Internally-driven implementation
- Externally-facilitated implementation (Experimental)
  Interventions: Behavioral: Externally-facilitated implementation

INTERVENTIONS:
Behavioral: Externally-facilitated implementation — NHs randomized to the externally-facilitated arm will attend the same kickoff meetings and have access to the same online resources as the control arm but will also be assigned a clinical coach and will have the opportunity to participate in a series of hosted peer-to-peer learning opportunities. The clinical coach will meet regularly with NH staff to guide the facility through implementation of the Wisconsin UTI Improvement Toolkit.
  Arms: Externally-facilitated implementation
Behavioral: Internally-driven implementation — Study NHs randomized to the control arm will participate in kickoff meetings introducing the different UTI toolkit components. The meeting will also cover topics on how to assemble a change team, how to use the different tools in the UTI toolkit, and how to track process and outcome measures to monitor progress. NHs assigned to the control arm will have access to a web-based data tracking tool that will allow them to trend a number of study outcomes (e.g., number of monthly urine cultures and UTI treatment events) in their facility over time. Instructions and educational tools will be made available as an online resource but otherwise NHs in the control arm will be expected to implement the Wisconsin UTI Improvement Toolkit using existing internal resources.
  Arms: Internally-driven implementation

SUMMARY:
The Wisconsin Healthcare-Associated Infections in Long-Term Care Coalition has developed a toolkit of evidence-based best practices to improve the management of urinary tract infection (UTI) in Wisconsin nursing homes (NHs). The theory and evidence supporting the individual improvement strategies promoted in the "Wisconsin UTI Improvement Toolkit" are strong but their combined impact on antibiotic prescribing in Wisconsin NHs is not known. Moreover, many Wisconsin NHs lack the internal resources and expertise to successfully implement and sustain the change interventions recommended in the toolkit. Consequently, there is a critical need to identify effective strategies to support implementation of best practices in this setting. The investigators hypothesize that an externally-facilitated implementation based on coaching and peer-to-peer learning will result in superior toolkit adoption and reduced rates of antibiotic utilization compared to a standard implementation.

To test these two hypotheses, the investigators are proposing a hybrid type 2 effectiveness-implementation randomized clinical trial in 20 Wisconsin NHs. Facilities randomized to the standard implementation approach will participate in a kickoff meeting and have access to a variety of online implementation resources. Facilities randomized to the enhanced implementation approach will have access to the same resources but will also be assigned a clinical coach and be invited to participate in ongoing collaborative learning sessions. The clinical coach will meet regularly with NH staff to guide the facility through implementation of the toolkit, including assembling a change team, performing an assessment to identify baseline barriers and facilitators of change, and ongoing integration of the toolkit practices into existing workflows. The learning collaborative will bring NH participants together to share change and improvement strategies with each other. UTI prescriptions per 1,000 resident-days in the study arms will be compared using generalized linear mixed models. A mixed methods evaluation structured around the REAIM framework (Reach, Effectiveness, Adoption, Implementation and Maintenance) will be employed to assess differences in toolkit implementation among facilities in both arms of the study.

ELIGIBILITY:
Criteria for Nursing Homes (Sample size 20)

Inclusion Criteria:

* Medicare and Medicaid (dually) certified nursing homes
* Long-term care and skilled nursing beds > 50 beds
* The management of the facility agrees to random allocation to control or intervention group
* The facility is able to submit 3 sequential months of data on facility urine culture and antibiotic treatment rates via the study web portal

Exclusion Criteria:

* Assisted living facility wards
* Specialty care (ventilator or strict rehabilitation) wards

Criteria for Nursing Home staff (for interviews and observations, sample size 400)

Inclusion Criteria:

For the interviews and observations, all facility-employed and per diem nursing staff (certified nursing assistants [CNA], licensed practical nurses [LPN] and registered nurses [RN]) who are responsible for the care of >3 residents will be included in the study. For the questionnaires, all nursing home clinical care staff will be invited to participate.

Exclusion Criteria:

For the interviews and observations, nursing home staff responsible for the care of at most 3 residents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 338 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2021-11-24 (Actual); Study Completion 2021-11-24 (Actual)

PRIMARY OUTCOMES:
Urine culture orders per 1,000 resident-days | Up to 12 months pre-implementation and up to 12 months post-implementation
Antibiotic starts for treatment of suspected UTI per 1,000 resident-days | Up to 12 months pre-implementation and up to 12 months post-implementation

SECONDARY OUTCOMES:
Days of therapy for treatment of suspected UTI per 1,000 resident-days | Up to 12 months pre-implementation and up to 12 months post-implementation
Fluoroquinolone antibiotic starts and days of therapy per 1000 resident-days | Up to 12 months pre-implementation and up to 12 months post-implementation
Percentage of antibiotic starts for UTI meeting appropriateness criteria | Up to 12 months pre-implementation and up to 12 months post-implementation
Percentage of urine cultures meeting appropriateness criteria | Up to 12 months pre-implementation and up to 12 months post-implementation
Percentage of urine cultures positive for resistant bacteria | Up to 12 months pre-implementation and up to 12 months post-implementation
Number of positive clostridium difficile tests | Up to 12 months pre-implementation and up to 12 months post-implementation
Number of transfers to hospitals or emergency departments per 1000 resident-days | Up to 12 months pre-implementation and up to 12 months post-implementation
Number of resident deaths per 1000 resident-days | Up to 12 months pre-implementation and up to 12 months post-implementation

CONTACTS AND LOCATIONS:
Overall Officials: Christopher J Crnich, MD, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin-Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ford JH 2nd, Nora AT, Crnich CJ. Moving behavioral interventions in nursing homes from planning to action: a work system evaluation of a urinary tract infection toolkit implementation. Implement Sci Commun. 2023 Dec 12;4(1):156. doi: 10.1186/s43058-023-00535-y. PMID 38087393
- [Derived] Ford JH 2nd, Vranas L, Coughlin D, Selle KM, Nordman-Oliveira S, Ryther B, Ewers T, Griffin VL, Eslinger A, Boero J, Hardgrove P, Crnich CJ. Effect of a Standard vs Enhanced Implementation Strategy to Improve Antibiotic Prescribing in Nursing Homes: A Trial Protocol of the Improving Management of Urinary Tract Infections in Nursing Institutions Through Facilitated Implementation (IMUNIFI) Study. JAMA Netw Open. 2019 Sep 4;2(9):e199526. doi: 10.1001/jamanetworkopen.2019.9526. PMID 31509204